CLINICAL TRIAL: NCT05430412
Title: Clinical Trial to Assess the Efficacy and Safety of Adding GMA to Infliximab in Paediatric Patients With Steroid-refractory Ulcerative Colitis
Brief Title: CT to Assess the Efficacy and Safety of Adding GMA to Infliximab in Paediatric Patients With Steroid-refractory Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adacyte Therapeutics SL (Industry)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUITAR
Record Dates: First submitted 2022-04-19; First posted 2022-06-24 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adacolumn (Experimental): Adacolumn is a non-pharmacological treatment which reduces the inflammation by removing specifically targeted white blood cells from the blood circulation. The Adacolumn is designed to be used in combination with the Adamonitor and its Adastand, and the Adacircuit. The column has a capacity of 335 mL and is filled with cellulose acetate beads of 2 mm in diameter as the column adsorptive leukocytapheresis carriers. The carriers are bathed in 130 mL of sterile saline until use when the column is primed with additional sterile saline and then with heparinized saline prior to use.
  Patients will receive 10 sessions with Adacolumn. It would be reduced between 5 - 10, according to the patient´s response and following PI valuation. Patients will receive Adacolumn with IFX for that period of time.
  Patients will have received previously IFX for 12-16 weeks. visits will be conducted every week, for the application of Adacolumn.
  Interventions: Device: Adacolumn

INTERVENTIONS:
Device: Adacolumn — The study will consist of 10 sessions of Adacolumn® treatment (once per week) and a follow-up period (from week 12 to week 40 since study inclusion).

SUMMARY:
The primary endpoint will be evaluated through the following variables: PUCAI score, IFX levels, and steroid treatment.

Clinical response to IFX will be evaluated through the PUCAI score. The response will be considered clinically significant if PUCAI points continue maintained below 30 during the study period. The IFX response will also be determined by IFX serum levels. A therapeutic IFX level, i.e. for achieving an adequate clinical response, is established above 6 μg/mL. Finally, the necessity, or not, of a steroid treatment during the study period will also be indicative of successful efficacy with GMA.

DETAILED DESCRIPTION:
The trial has the following objectives:

Primary objective (PO):

The primary endpoint will be evaluated through the following variables: PUCAI score, IFX levels, and steroid treatment.

Clinical response to IFX will be evaluated through the PUCAI score. The response will be considered clinically significant if PUCAI points continue maintained below 30 during the study period. The IFX response will also be determined by IFX serum levels. A therapeutic IFX level, i.e. for achieving an adequate clinical response, is established above 6 μg/mL. Finally, the necessity, or not, of a steroid treatment during the study period will also be indicative of successful efficacy with GMA.

Secondary objectives (SO):

1. Quantification of IFX trough and ATI levels, and description of the IFX dose at baseline, 12 and 40 weeks of follow-up.
2. Measurement of PUCAI score at baseline, 12 and 40 weeks of follow-up.
3. Patients maintaining clinical response off steroids, 12 and 40 weeks of follow-up.
4. Patients experiencing flares-ups during the study period.
5. Quantification of fecal calprotectin level at baseline, 12 and 40 weeks of follow-up. Fecal calprotectin is associated with clinical remission with levels higher than 150 μg/g.
6. Measurement of C-reactive protein, erythrocyte sedimentation rate, hemoglobin, albumin, platelet levels at baseline, 12 and 40weeks of follow-up.
7. Quantification of leucocyte counts in peripheral blood at baseline, 12 and 40 weeks of followup.
8. Monitoring of AEs during the study period

ELIGIBILITY:
Inclusion Criteria:

1. Patients under 18 years of age and weighing ≥25 kg at the time of study initiation.
2. Patients with diagnosis of UC.
3. Patients who started IFX treatment due to the lack of response to corticosteroids following an UC flare-up (steroid-refractory UC).
4. Patients who have received IFX between 12 and 16 weeks prior to the study initiation.
5. Patients who have showed a clinical response to IFX at the time of study initiation (defined as a reduction of at least 15 points in PUCAI score and being maintained below 30 points).
6. Patients with therapeutic IFX blood levels (above 6 μg/mL) at the time of study initiation.
7. Patient´s legal guardian must be willing and able to give written informed consent, and the patient must be willing to give written informed assent (if applicable as determined by the Ethics Committee) and comply with the Study visit Schedule.

Exclusion Criteria:

1. Patients who have received another anti-TNF prior to entry in the study.
2. Patients with a peripheral circulation count of less than 2,000 granulocytes per μL.
3. Pregnant and lactating of childbearing potential patients.
4. Participation in another study or use of any experimental therapy within 30 days before day 1 of Study initiation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary objective:evaluate if Adacolumn® can sustain clinical response to IFX for 12 weeks of follow-up (V.11) or 40 weeks of follow-up (V18). Clinical response to IFX will be evaluated through PUCAI SCORE | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of PUCAI score as continuous variable at V.11 and at V.18 will be performed. Response to IFX will be clinically significant if PUCAI score continues maintained below 30 during the study (follow-up visits), so the nº and % of patients with a PUCAI score below 30 points in all visits between baseline to V.11 and baseline to V.18 will be described. Furthermore, comparison scores in both visits (baseline vs. V.11 and baseline vs. V.18) will be performed, by means of absolute and relative changes
Primary objective: evaluate if Adacolumn® can sustain clinical response to IFX for 12 weeks of follow-up (V.11) or 40 weeks of follow-up (V18). Clinical response to IFX will be evaluated through IFX-LEVELS | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of IFX levels as continuous variable at V.11 and at V.18 will be performed. Response to IFX will be clinically significant if IFX levels > 6 μg/mL during the study, so the nº and % of patients with a IFX level > 6 μg/mL in all visits between baseline to V.11 and baseline to V.18 will be described. Furthermore, comparison between IFX levels in both visits will be performed, by means of absolute and relative changes
Primary objective:evaluate if Adacolumn® can sustain clinical response to IFX for 12 weeks of follow-up (V.11) or 40 weeks of follow-up (V18). Clinical response to IFX will be evaluated through STEROIDS USE | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of the number and percentage of patients with a change in steroids treatment from baseline to V.11 and from baseline to V.18. Furthermore, comparison between visits will be performed.

SECONDARY OUTCOMES:
To evaluate the IFX and ATI level variations in the treatment regimen during the study period. Quantification of IFX trough and ATI levels, and description of the IFX dose at baseline, 12 and 40 weeks of follow-up | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of IFX blood and ATI levels as continuous variables at baseline visit, Visit 11 (12 weeks) and Visit 18 (40 weeks) will be performed. Their variation between visits (baseline vs. Visit 11 and baseline vs. Visit 18) will be analysed by means of absolute and relative change. Moreover, description of IFX dose by kilogram will be described in these visits
To measure the PUCAI score variation during the study period. Measurement of PUCAI score at baseline, 12 and 40 weeks of follow-up. | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of PUCAI score as continuous variable at baseline visit, Visit 11 (12 weeks) and Visit 18 (40 weeks) will be performed. Its variation between visits (baseline vs. Visit 11 and baseline vs. Visit 18) will be analysed by means of absolute and relative change
To determine the percentage of patients maintaining steroid-free response during the study period at 12 and 40 weeks. | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of the number and percentage of patients changing the behaviour of steroids treatment (use or not use) from baseline visit to Visit 11 (12 weeks) and from baseline visit to Visit 18 (40 weeks) will be computed. Furthermore, comparison between visits (baseline vs. Visit 11 and baseline vs. Visit 18) will be performed
To describe the number of flare-ups during the study period. Patients experiencing flares-ups during the study period. | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of the number of patients experienced flare-ups and the accumulate number of flare-ups from baseline visit to Visit 11 and from baseline visit to Visit 18 will be computed.
To measure faecal calprotectin level during the study period. Quantification of faecal calprotectin level at baseline, 12 and 40 weeks of follow-up. Faecal calprotectin is associated with clinical remission with levels higher than 150 μg/g. | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of faecal calprotectin level as continuous variable at baseline visit, Visit 11 (12 weeks) and Visit 18 (40 weeks) will be performed. Their variation between visits (baseline vs. Visit 11 and baseline vs. Visit 18) will be analysed by means of absolute and relative change. As levels of faecal calprotectin > 150 μg/g are associated with clinical remission, the number and percentage of patients with faecal calprotectin > 150 μg/g will be described. Furthermore, comparison between visits (baseline vs. Visit 11 and baseline vs. Visit 18) will be performed.
To monitor the evolution of biochemical markers of inflammatory activity in UC and other laboratory parameters. Measurement of C-reactive protein, ESR, haemoglobin, albumin, platelet levels, PT, granulocytes at baseline, 12(V11) and 40 weeks(V18) | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of CRP, ESR, haemoglobin, albumin platelet levels, PT and granulocytes as continuous variables at baseline visit, Visit 11 (12 weeks) and Visit 18 (40 weeks) will be performed. Their variation between visits (baseline vs. Visit 11 and baseline vs. Visit 18) will be analysed by means of absolute and relative change.
To determine the evolution of leucocyte counts in peripheral blood during the study period. Quantification of leucocyte counts in peripheral blood at baseline, 12 and 40 weeks of follow-up. | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  Description of leucocyte counts as continuous variable at Baseline visit, Visit 11 (12 weeks) and Visit 18 (40 weeks) will be performed. Its variation between visits (baseline vs. Visit 11 and baseline vs. Visit 18) will be analysed by means of absolute and relative change
To evaluate the safety of Adacolumn® during the study period, all the recorded AEs will be described by: | Baseline visit vs Visit 11 (12 weeks) (interim analysis). Baseline visit vs Visit 18 (40 weeks) (for final analysis)
  * The number of patients who suffer them
  * The number of patients who suffer AEs related to Adacolumn®
  * Their incidence and duration
  * Their relationship with Adacolumn®
  * Seriousness, severity, ongoing and outcome This analysis will be done on those patients belonging to the safety sample

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Martín de Carpi, Study Chair — Hospital San Joan de Deu; Jorge Manuel Bastos Amil Dias, Study Chair — CHU Sao Joao
Locations (10):
- Portugal (3):
  - Hospital Coimbra, Coimbra
  - Hospital Santa Maria, Lisbon
  - Hospital Soa Joao, Porto
- Spain (7):
  - Hospital H. Sant Joan de Déu, Sant Joan Despí, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Materno-Infantil del H.U.R. de Málaga, Málaga
  - Hospital U. Ntra Señora de Candelaria, Santa Cruz de Tenerife
  - Complejo H. Regional Virgen Del Rocío, Seville
  - Hospital Universitari I Politècnic La Fe, Valencia

REFERENCES:
- [Background] Saniabadi AR, Hanai H, Takeuchi K, Umemura K, Nakashima M, Adachi T, Shima C, Bjarnason I, Lofberg R. Adacolumn, an adsorptive carrier based granulocyte and monocyte apheresis device for the treatment of inflammatory and refractory diseases associated with leukocytes. Ther Apher Dial. 2003 Feb;7(1):48-59. doi: 10.1046/j.1526-0968.2003.00012.x. PMID 12921115
- [Background] Shimoyama T, Sawada K, Hiwatashi N, Sawada T, Matsueda K, Munakata A, Asakura H, Tanaka T, Kasukawa R, Kimura K, Suzuki Y, Nagamachi Y, Muto T, Nagawa H, Iizuka B, Baba S, Nasu M, Kataoka T, Kashiwagi N, Saniabadi AR. Safety and efficacy of granulocyte and monocyte adsorption apheresis in patients with active ulcerative colitis: a multicenter study. J Clin Apher. 2001;16(1):1-9. doi: 10.1002/jca.1000. PMID 11309823
- [Background] Saniabadi AR, Tanaka T, Yamamoto T, Kruis W, Sacco R. Granulomonocytapheresis as a cell-dependent treatment option for patients with inflammatory bowel disease: Concepts and clinical features for better therapeutic outcomes. J Clin Apher. 2019 Feb;34(1):51-60. doi: 10.1002/jca.21670. Epub 2018 Nov 8. PMID 30407662
- [Background] Yoshimura N, Tadami T, Kawaguchi T, Sako M, Yoshimoto H, Yamaka T, Takazoe M. Processed blood volume impacts clinical efficacy in patients with ulcerative colitis undergoing adsorptive depletion of myeloid lineage leucocytes. J Gastroenterol. 2012 Jan;47(1):49-55. doi: 10.1007/s00535-011-0464-0. Epub 2011 Sep 14. PMID 21915624
- [Background] Suzuki Y, Yoshimura N, Saniabadi AR, Saito Y. Selective granulocyte and monocyte adsorptive apheresis as a first-line treatment for steroid naive patients with active ulcerative colitis: a prospective uncontrolled study. Dig Dis Sci. 2004 Apr;49(4):565-71. doi: 10.1023/b:ddas.0000026299.43792.ae. PMID 15185858
- [Background] Suzuki Y, Yoshimura N, Fukuda K, Shirai K, Saito Y, Saniabadi AR. A retrospective search for predictors of clinical response to selective granulocyte and monocyte apheresis in patients with ulcerative colitis. Dig Dis Sci. 2006 Nov;51(11):2031-8. doi: 10.1007/s10620-006-9199-9. Epub 2006 Sep 27. PMID 17004123
- [Background] Hanai H, Watanabe F, Takeuchi K, Iida T, Yamada M, Iwaoka Y, Saniabadi A, Matsushita I, Sato Y, Tozawa K, Arai H, Furuta T, Sugimoto K, Bjarnason I. Leukocyte adsorptive apheresis for the treatment of active ulcerative colitis: a prospective, uncontrolled, pilot study. Clin Gastroenterol Hepatol. 2003 Jan;1(1):28-35. doi: 10.1053/jcgh.2003.50005. PMID 15017514
- [Background] Saez-Gonzalez E, Moret I, Alvarez-Sotomayor D, Diaz-Jaime FC, Cerrillo E, Iborra M, Nos P, Beltran B. Immunological Mechanisms of Adsorptive Cytapheresis in Inflammatory Bowel Disease. Dig Dis Sci. 2017 Jun;62(6):1417-1425. doi: 10.1007/s10620-017-4577-z. Epub 2017 Apr 21. PMID 28432476
- [Background] Dignass A, Akbar A, Hart A, Subramanian S, Bommelaer G, Baumgart DC, Grimaud JC, Cadiot G, Makins R, Hoque S, Bouguen G, Bonaz B. Safety and Efficacy of Granulocyte/Monocyte Apheresis in Steroid-Dependent Active Ulcerative Colitis with Insufficient Response or Intolerance to Immunosuppressants and/or Biologics [the ART Trial]: 12-week Interim Results. J Crohns Colitis. 2016 Jul;10(7):812-20. doi: 10.1093/ecco-jcc/jjw032. Epub 2016 Jan 27. PMID 26818659
- [Background] Dignass A, Akbar A, Baumgart DC, Bommelaer G, Bouguen G, Cadiot G, Gillessen A, Grimaud JC, Hart A, Hoque S, Makins R, Michiels C, Moreau J, Premchand P, Ramlow W, Schanz S, Subramanian S, von Tirpitz C, Bonaz B. Granulocyte/monocyte adsorptive apheresis for the treatment of therapy-refractory chronic active ulcerative colitis. Scand J Gastroenterol. 2018 Apr;53(4):442-448. doi: 10.1080/00365521.2018.1447598. Epub 2018 Mar 7. PMID 29513111
- [Background] Martin de Carpi J, Vilar P, Prieto G, Garcia Novo MD, Ribes C, Varea V. Safety and efficacy of granulocyte and monocyte adsorption apheresis in paediatric inflammatory bowel disease: a prospective pilot study. J Pediatr Gastroenterol Nutr. 2008 Apr;46(4):386-91. doi: 10.1097/MPG.0b013e31815604e5. PMID 18367949
- [Background] Ruuska T, Kuster P, Grahnquist L, Lindgren F, Wewer AV. Efficacy and safety of granulocyte, monocyte/macrophage adsorptive in pediatric ulcerative colitis. World J Gastroenterol. 2016 May 7;22(17):4389-96. doi: 10.3748/wjg.v22.i17.4389. PMID 27158208
- [Background] Golbabapour S, da Silva LM, Athanasiou A. Immunological Aspects of Gastrointestinal Diseases. Gastroenterol Res Pract. 2017;2017:2891574. doi: 10.1155/2017/2891574. Epub 2017 May 17. No abstract available. PMID 28620414
- [Background] Ghosh S, Shand A, Ferguson A. Ulcerative colitis. BMJ. 2000 Apr 22;320(7242):1119-23. doi: 10.1136/bmj.320.7242.1119. No abstract available. PMID 10775225
- [Background] Nedelciuc O, Pintilie I, Dranga M, Mihai C, Prelipcean CC. Quality of life in patients with ulcerative colitis. Rev Med Chir Soc Med Nat Iasi. 2012 Jul-Sep;116(3):756-60. PMID 23272523
- [Background] Ruemmele FM, Hyams JS, Otley A, Griffiths A, Kolho KL, Dias JA, Levine A, Escher JC, Taminiau J, Veres G, Colombel JF, Vermeire S, Wilson DC, Turner D. Outcome measures for clinical trials in paediatric IBD: an evidence-based, expert-driven practical statement paper of the paediatric ECCO committee. Gut. 2015 Mar;64(3):438-46. doi: 10.1136/gutjnl-2014-307008. Epub 2014 May 12. PMID 24821616
- [Background] Tanaka T, Yamamoto T, Sawada K, Sacco R. Treatment options for children and adolescents with inflammatory bowel disease: is granulomonocytapheresis an effective alternative to drug therapy? Expert Rev Gastroenterol Hepatol. 2017 Aug;11(8):749-758. doi: 10.1080/17474124.2017.1341309. Epub 2017 Jun 28. PMID 28612637
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Roda G, Jharap B, Neeraj N, Colombel JF. Loss of Response to Anti-TNFs: Definition, Epidemiology, and Management. Clin Transl Gastroenterol. 2016 Jan 7;7(1):e135. doi: 10.1038/ctg.2015.63. PMID 26741065
- [Background] Zitomersky NL, Atkinson BJ, Fournier K, Mitchell PD, Stern JB, Butler MC, Ashworth L, Hauenstein S, Heiner L, Chuang E, Singh S, Bousvaros A. Antibodies to infliximab are associated with lower infliximab levels and increased likelihood of surgery in pediatric IBD. Inflamm Bowel Dis. 2015 Feb;21(2):307-14. doi: 10.1097/MIB.0000000000000284. PMID 25569737
- [Background] Thanaraj S, Hamlin PJ, Ford AC. Systematic review: granulocyte/monocyte adsorptive apheresis for ulcerative colitis. Aliment Pharmacol Ther. 2010 Dec;32(11-12):1297-306. doi: 10.1111/j.1365-2036.2010.04490.x. Epub 2010 Oct 14. PMID 21050231
- [Background] Rolandsdotter H, Eberhardson M, Fagerberg UL, Finkel Y. Granulocyte and Monocyte Apheresis for Induction of Remission in Children With New-Onset Inflammatory Bowel Colitis. J Pediatr Gastroenterol Nutr. 2018 Jan;66(1):84-89. doi: 10.1097/MPG.0000000000001641. PMID 28604509
- [Background] Yamamoto T, Umegae S, Matsumoto K. Long-term clinical impact of early introduction of granulocyte and monocyte adsorptive apheresis in new onset, moderately active, extensive ulcerative colitis. J Crohns Colitis. 2012 Aug;6(7):750-5. doi: 10.1016/j.crohns.2011.12.009. Epub 2012 Jan 12. PMID 22398094
- [Background] Yokoyama Y, Sawada K, Aoyama N, Yoshimura N, Sako M, Hirai F, Kashiwagi N, Suzuki Y. Efficacy of Granulocyte and Monocyte Adsorptive Apheresis in Patients With Inflammatory Bowel Disease Showing Lost Response to Infliximab. J Crohns Colitis. 2020 Sep 16;14(9):1264-1273. doi: 10.1093/ecco-jcc/jjaa051. PMID 32166331
- [Background] Rodriguez-Lago I, Sempere L, Gutierrez A, Nunez A, Leo Carnerero E, Hinojosa E, Mora M, Canete F, Manosa M, Herrera C, Beltran B, Fores A, Arjona D, Barreiro-de Acosta M, Khorrami S, Aguirre U, Ginard D, Cabriada JL. Granulocyte-monocyte apheresis: an alternative combination therapy after loss of response to anti-TNF agents in ulcerative colitis. Scand J Gastroenterol. 2019 Apr;54(4):459-464. doi: 10.1080/00365521.2019.1600715. Epub 2019 Apr 14. PMID 30982369
- [Background] Yokoyama Y, Kamikozuru K, Watanabe K, Nakamura S. Inflammatory bowel disease patients experiencing a loss of response to infliximab regain long-term response after undergoing granulocyte/monocyte apheresis: A case series. Cytokine. 2018 Mar;103:25-28. doi: 10.1016/j.cyto.2017.12.030. Epub 2017 Dec 29. PMID 29291447
- [Background] Velasco Rodriguez-Belvis M, Viada Bris JF, Palomino Perez L, Munoz Codoceo RA. Regain of Response to Adalimumab in a Steroid-Dependent Pediatric Patient With Ulcerative Colitis After Undergoing Selective Granulocyte and Monocyte Apheresis. Inflamm Bowel Dis. 2019 Jun 18;25(7):e82-e83. doi: 10.1093/ibd/izy404. No abstract available. PMID 30698787
- [Background] Saniabadi AR, Hanai H, Suzuki Y, Ohmori T, Sawada K, Yoshimura N, Saito Y, Takeda Y, Umemura K, Kondo K, Ikeda Y, Fukunaga K, Nakashima M, Beretta A, Bjarnason I, Lofberg R. Adacolumn for selective leukocytapheresis as a non-pharmacological treatment for patients with disorders of the immune system: an adjunct or an alternative to drug therapy? J Clin Apher. 2005 Oct;20(3):171-84. doi: 10.1002/jca.20046. PMID 15892107
- [Background] Turner D, Otley AR, Mack D, Hyams J, de Bruijne J, Uusoue K, Walters TD, Zachos M, Mamula P, Beaton DE, Steinhart AH, Griffiths AM. Development, validation, and evaluation of a pediatric ulcerative colitis activity index: a prospective multicenter study. Gastroenterology. 2007 Aug;133(2):423-32. doi: 10.1053/j.gastro.2007.05.029. Epub 2007 May 21. PMID 17681163
- [Background] Dotson JL, Crandall WV, Zhang P, Forrest CB, Bailey LC, Colletti RB, Kappelman MD. Feasibility and validity of the pediatric ulcerative colitis activity index in routine clinical practice. J Pediatr Gastroenterol Nutr. 2015 Feb;60(2):200-4. doi: 10.1097/MPG.0000000000000568. PMID 25221935
- [Background] Ungar B, Levy I, Yavne Y, Yavzori M, Picard O, Fudim E, Loebstein R, Chowers Y, Eliakim R, Kopylov U, Ben-Horin S. Optimizing Anti-TNF-alpha Therapy: Serum Levels of Infliximab and Adalimumab Are Associated With Mucosal Healing in Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2016 Apr;14(4):550-557.e2. doi: 10.1016/j.cgh.2015.10.025. Epub 2015 Oct 29. PMID 26538204
- [Background] Measurement of infliximab and anti-infliximab antibody levels can help distinguish maintenance versus loss of response. Gastroenterol Hepatol (N Y). 2012 Feb;8(2):131-4. No abstract available. PMID 22485082
- [Background] Costa F, Mumolo MG, Ceccarelli L, Bellini M, Romano MR, Sterpi C, Ricchiuti A, Marchi S, Bottai M. Calprotectin is a stronger predictive marker of relapse in ulcerative colitis than in Crohn's disease. Gut. 2005 Mar;54(3):364-8. doi: 10.1136/gut.2004.043406. PMID 15710984
- [Background] Rodriguez-Lago I, Gomez-Irwin L, Fernandez E, Higuera R, Cabriada JL. Granulocyte-Monocyte Apheresis as an Adjuvant Therapy to Anti-Tumor Necrosis Factor Drugs for Ulcerative Colitis. Ther Apher Dial. 2017 Feb;21(1):26-30. doi: 10.1111/1744-9987.12485. Epub 2017 Jan 11. PMID 28078747
- [Background] Turner D, Ruemmele FM, Orlanski-Meyer E, Griffiths AM, de Carpi JM, Bronsky J, Veres G, Aloi M, Strisciuglio C, Braegger CP, Assa A, Romano C, Hussey S, Stanton M, Pakarinen M, de Ridder L, Katsanos K, Croft N, Navas-Lopez V, Wilson DC, Lawrence S, Russell RK. Management of Paediatric Ulcerative Colitis, Part 1: Ambulatory Care-An Evidence-based Guideline From European Crohn's and Colitis Organization and European Society of Paediatric Gastroenterology, Hepatology and Nutrition. J Pediatr Gastroenterol Nutr. 2018 Aug;67(2):257-291. doi: 10.1097/MPG.0000000000002035. PMID 30044357
- [Background] Zhu M, Xu X, Nie F, Tong J, Xiao S, Ran Z. The efficacy and safety of selective leukocytapheresis in the treatment of ulcerative colitis: a meta-analysis. Int J Colorectal Dis. 2011 Aug;26(8):999-1007. doi: 10.1007/s00384-011-1193-9. Epub 2011 Apr 8. PMID 21476027
- See also: Adacyte Therapeutics Therapeutics. Adacolumn®. Instructions for use — https://www.adacyte.com/professional/products/adacolumn/
- See also: Adacyte Therapeutics — https://www.adacyte.com
- See also: European Commission. Ethical Considerations for Clinical Trials — https://ec.europa.eu/health/sites/health/files/files/eudralex/vol-10/ethical_considerations_en.pdf
- See also: European Medicines Agency. Informed Consent for Paediatric Clinical Trials in Europe 2015 — https://www.ema.europa.eu/en/documents/other/informed-consent-paediatric-clinical-trials-europe-2015_en.pdf